CLINICAL TRIAL: NCT03105102
Title: A Multicenter, Randomized, Double-Blind, Placebo Controlled 52-Week Maintenance and an Open-Label Extension Study of the Efficacy and Safety of Risankizumab in Subjects With Crohn's Disease
Brief Title: A Study of the Efficacy and Safety of Risankizumab in Participants With Crohn's Disease
Acronym: FORTIFY
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-000; 2023-506399-28-00 (Other: EU CT)
Expanded Access: Available
Record Dates: First submitted 2017-04-04; First posted 2017-04-07 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease
Keywords: Risankizumab; ABBV-066; BI 655066; SKYRIZI; Crohn's Disease (CD)
MeSH Terms: conditions — Crohn Disease | interventions — risankizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Double-blind Placebo for Risankizumab (Sub-Study 1) (Placebo Comparator): Participants randomized to receive double-blind placebo for risankizumab for 52 weeks.
  Interventions: Drug: Placebo for Risankizumab SC
- Double-blind Risankizumab Dose 1 (Sub-Study 1) (Experimental): Participants randomized to receive double-blind risankizumab dose 1 for 52 weeks.
  Interventions: Drug: Risankizumab SC
- Double-blind Risankizumab Dose 2 (Sub-Study 1) (Experimental): Participants randomized to receive double-blind risankizumab dose 2 for 52 weeks.
  Interventions: Drug: Risankizumab SC
- Maintenance Risankizumab Dose 1 (Sub-Study 2) (Experimental): Participants will receive double-blind subcutaneous (SC)risankizumab dose 1 and intravenous placebo at Week 0 followed by open-label SC risankizumab dose 1 from Week 8 through Week 52.
  Interventions: Drug: Placebo for Risankizumab IV; Drug: Risankizumab SC
- Maintenance Risankizumab Dose 2 (Sub-Study 2) (Experimental): Participants will receive double-blind subcutaneous placebo and intravenous risankizumab dose 3 at Week 0 followed by open-label SC risankizumab dose 1 from Week 8 through Week 52.
  Interventions: Drug: Placebo for Risankizumab SC; Drug: Risankizumab IV; Drug: Risankizumab SC
- Open-label Risankizumab (Sub-Study 3) (Experimental): Participants who completed Sub-study 1 or Sub-study 2 or other AbbVie risankizumab Crohn's disease study or M16-006 or M15-991 without endoscopy will receive open-label risankizumab dose 1 or dose 2 depending on their preceding study beginning at Week 56.
  Interventions: Drug: Risankizumab SC
- Risankizumab On-Body Injector and Open Label (Sub-Study 4) (Experimental): Participants in Sub-study 3 who meet eligible criteria for Sub-study 4 will receive risankizumab dose 1 or dose 2 via on-body injectors on Weeks 0,8 and 16. Beginning Week 24, participants will receive risankizumab dose 1 or dose 2 via pre-filled syringes Q8W.
  Interventions: Drug: Risankizumab SC; Drug: Risankizumab On-Body Injector (OBI)
- CTE: Open Label Continuous Treatment Extension (Experimental): Participants who tolerate and derive benefit from receiving risankizumab and complete Sub-study 3 or Sub-study 4 will receive risankizumab dose 1 or dose 2 Q8W.
  Interventions: Drug: Risankizumab SC

INTERVENTIONS:
Drug: Placebo for Risankizumab SC — Placebo for Risankizumab SC Subcutaneous (SC) Injection
  Arms: Double-blind Placebo for Risankizumab (Sub-Study 1); Maintenance Risankizumab Dose 2 (Sub-Study 2)
Drug: Risankizumab IV — Risankizumab IV Intravenous (IV) infusion
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Maintenance Risankizumab Dose 2 (Sub-Study 2)
Drug: Placebo for Risankizumab IV — Placebo for Risankizumab IV Intravenous (IV) infusion
  Arms: Maintenance Risankizumab Dose 1 (Sub-Study 2)
Drug: Risankizumab SC — Risankizumab SC Subcutaneous (SC) injection
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: CTE: Open Label Continuous Treatment Extension; Double-blind Risankizumab Dose 1 (Sub-Study 1); Double-blind Risankizumab Dose 2 (Sub-Study 1); Maintenance Risankizumab Dose 1 (Sub-Study 2); Maintenance Risankizumab Dose 2 (Sub-Study 2); Open-label Risankizumab (Sub-Study 3); Risankizumab On-Body Injector and Open Label (Sub-Study 4)
Drug: Risankizumab On-Body Injector (OBI) — Subcutaneous (SC) injection; on-body injector (OBI)
  Other Names: ABBV-066; BI 655066; SKYRIZI
  Arms: Risankizumab On-Body Injector and Open Label (Sub-Study 4)

SUMMARY:
The study consists of 4 sub-studies, as follows:

* Sub-study 1 (Randomized, double-blind, placebo controlled study) to evaluate the efficacy and safety of risankizumab versus placebo as maintenance therapy in participants with moderately to severely active Crohn's disease (CD) who responded to intravenous risankizumab induction treatment in Study M16-006 or Study M15-991;
* Sub-study 2 (Randomized, exploratory maintenance study) to evaluate the efficacy and safety of two different dosing regimens for risankizumab as maintenance therapy in participants who responded to induction treatment in Study M16-006 or Study M15-991;
* Sub-study 3 (Open-label, long-term extension study) to evaluate long-term safety of risankizumab in participants who completed Sub-study 1, Sub-study 2, another AbbVie risankizumab Crohn's disease study, or participants who responded to induction treatment in Study M16-006 or Study M15-991 with no final endoscopy due to the Covid-19 pandemic. Additional objectives are to further investigate long-term efficacy and tolerability of risankizumab;
* Sub-study 4 (Open-label On Body Injector (OBI) administration and long-term extension study) to evaluate patient-reported outcomes, efficacy, safety, tolerability, and pharmacokinetics of risankizumab administered via OBI in participants who are receiving maintenance treatment with risankizumab.
* OL CTE to ensure uninterrupted care in accordance with local regulations until risankizumab is commercially available for participants who completed Sub-study 3, Sub-study 4.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have entered and completed Study M16-006 or Study M15-991 or other AbbVie risankizumab Crohn's disease study.
* Participants have completed the study M16-006 or M15-991 and have achieved clinical response.
* Sub-Study 4:

  * Participants receiving maintenance treatment in Sub-study 3 and willing to comply with the requirements of Sub-study 4, including self-administration of sub-cutaneous injections using the on-body injector (OBI).
  * Participant has received at least 16 weeks of stable dosing with risankizumab in Sub-study 3 (i.e., no rescue within 16 weeks and participant has surpassed the 72-week mark).

Exclusion Criteria:

* Participants should not be enrolled in Study M16-000 with high grade colonic dysplasia or colon cancer identified during Study M15-991, Study M16-006 or another AbbVie risankizumab Crohn's disease study if the final endoscopy was performed prior to enter Study M16-000 OR is considered by the Investigator, for any reason, to be an unsuitable candidate for the study.
* Participant who has a known hypersensitivity to risankizumab or the excipients of any of the study drugs or the ingredients of Chinese hamster ovary (CHO), OR had an adverse event (AE) during Studies M16-006, M15-991 or another AbbVie risankizumab Crohn's disease study that in the Investigator's judgment makes the participant unsuitable for this study.
* Participant is not in compliance with prior and concomitant medication requirements throughout Studies M16-006, M15-991 or another AbbVie risankizumab Crohn's disease study.
* Confirmed positive urine pregnancy test at the Final Visit of Study M16-006, Study M15-991 or another AbbVie risankizumab Crohn's disease study.
* Have a known history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease, such as lymphadenopathy and/or splenomegaly.
* Any active or chronic recurring infections based on the Investigator's assessment makes the participant an unsuitable candidate for the study.

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1336 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Sub-Study 1: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission | Week 52
  The CDAI is used to evaluate disease activity in patients with Crohn's disease. The CDAI clinical remission is defined as a CDAI score of < 150.
Sub-Study 1: Percentage of Participants With Endoscopic Response | Week 52
  Endoscopic response defined as decrease from Baseline of the induction study in Simple Endoscopic Score for Crohn's Disease (SES-CD).
Sub-Study 3: Number of Participants With Adverse Events | Up to Week 220
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. The investigator assessed the relationship of each event to the use of study drug as either probably related, possibly related, probably not related or not related. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the subject and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent AEs are defined as any event that began or worsened in severity after the first dose of study drug. For more details on adverse events please see the Adverse Event section.
Sub-Study 4: Percentage of Participants With an Observer Rating of Successful Participant Self Administration | Up to Week 16
  Participant who successfully completed the sequence of critical steps in the instructions for use (IFU) without errors to administer study drug via the OBI at Week 0 and 16.
Sub-Study 4: Percentage of Participants who had no Potential Hazards | Up to Week 16
  Measured by an observer on the possible use-related hazards checklist for self-administration with OBI at Week 0 and Week 16.
Sub-Study 4: Percentage of Participants Rating of Acceptability Using Self-Injection Assessment Questionnaire (SIAQ) at Weeks 0, 8, 16 | Up to Week 16
  SIAQ evaluations consist of the PRE module, which is self-completed immediately before the first OBI self-injection at baseline, and the POST module, which is self-completed 20 to 40 min following injections at Weeks 0, 8, 16. These modules are completed by participants while alone in a quiet environment.
  Participants rate each item of the SIAQ. The ratings are later transformed to scores ranging from 0 (worst experience) to 10 (best experience). The domain score is the mean of the item scores included in the domain. Domain scores are calculated only if at least half of the domain items are completed. Item and domain scores from the PRE module are compared with the corresponding item and domain scores from the POST modules.
Sub-Study 4: Percentage of Participants in CDAI Clinical Remission at Week 0, 16 | Up to Week 16
  Clinical remission per average daily stool frequency (SF) and average daily abdominal pain (AP) score.

SECONDARY OUTCOMES:
Sub-Study 1: Percentage of Participants With Clinical Remission | Week 52
  Clinical remission per average daily stool frequency (SF) and average daily AP score.
Sub-Study 1: Percentage of Participants With CDAI Clinical Remission Among Participants With CDAI Clinical Remission in Week 0 | Week 52
  The CDAI is used to evaluate disease activity in patients with Crohn's disease
Sub-Study 1: Percentage of Participants With Ulcer-Free Endoscopy | Week 52
  Endoscopic healing was assessed using SES-CD.
Sub-Study 1: Percentage of Participants With Endoscopic Remission | Week 52
  Endoscopic Remission is defined as SES-CD <= 4 and at least a 2 point reduction versus baseline and no subscore greater than 1 in any individual variable, as scored by a central reviewer
Sub-Study 1: Change From Baseline of Induction in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) | Week 52
  The FACIT-Fatigue is a validated tool that measures an individual's level of fatigue during their usual daily activities over the past week.
Sub-Study 1: Percentage of Participants Who Discontinued Corticosteroid Use for 90 Days and Achieved Clinical Remission in Participants Taking Steroids at Baseline | Week 52
  Participants who discontinued corticosteroid use and achieved clinical remission per average daily SF and average daily AP score.
Sub-Study 1: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Response | Week 52
  The CDAI is used to evaluate disease activity in patients with Crohn's disease.
Sub-Study 1: Percentage of Participants With Stool Frequency (SF) Remission | Week 52
  SF Remission is defined by an average daily SF <= 2.8 and not worse than baseline.
Sub-Study 1: Percentage of Participants With Abdominal Pain (AP) Remission | Week 52
  AP Remission is defined by an average daily AP <= 1 and not worse than baseline.
Sub-Study 1: Percentage of Participants With CDAI Clinical Remission and Endoscopic Response | Week 52
  The CDAI is used to evaluate disease activity in patients with Crohn's disease. The CDAI clinical remission is defined as a CDAI score of < 150. Endoscopic response defined as decrease from baseline of > 50% of the induction study in Simple Endoscopic Score for Crohn's Disease (SES-CD).
Sub-Study 1: Percentage of Participants With Deep Remission | Week 52
  Deep remission defined as participants with both clinical remission (per average daily SF and average daily AP score) and endoscopic remission (assessed using SES-CD).
Sub-Study 1: Percentage of Participants With Exposure Adjusted Occurrence of CD-related Hospitalizations From Week 0 Through Week 52 | Up to Week 52
  Participants with an event that results in admission to the hospital.

OTHER OUTCOMES:
Sub-Study 2: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Clinical Remission | Week 52
  The CDAI is used to evaluate disease activity in patients with Crohn's disease. The CDAI clinical remission is defined as a CDAI score of < 150.
Sub-Study 2: Percentage of Participants With Endoscopic Response | Week 52
  Endoscopic response defined as decrease from Baseline of the induction study in Simple Endoscopic Score for Crohn's Disease (SES-CD).
Sub-Study 2: Percentage of Participants With Exposure Adjusted Occurrence of CD-related Hospitalizations From Week 0 Through Week 52 | Up to Week 52
  Participants with an event that results in admission to the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (496):
- United States (111):
  - Digestive Disease Consultants, A Division of Arizona Digestive Health, P.C /ID# 211884, Mesa, Arizona
  - Phoenix VA Health Care System /ID# 162264, Phoenix, Arizona
  - Banner - University Medical Center Tucson /ID# 158502, Tucson, Arizona
  - Atria Clinical Research /ID# 164505, Little Rock, Arkansas
  - Southern California Res. Ctr. /ID# 211991, Coronado, California
  - Duplicate_Newport Huntington Medical Group /ID# 213035, Huntington Beach, California
  - UC San Diego Health Systems /ID# 155555, La Jolla, California
  - United Medical Doctors /ID# 207888, Los Alamitos, California
  - TLC Clinical Research Inc /ID# 212719, Los Angeles, California
  - Gastrointestinal Biosciences Clinical Trials, LLC /ID# 162657, Los Angeles, California
  - United Medical Doctors - Murrieta /ID# 158300, Murrieta, California
  - University of California San Francisco - Mission Bay /ID# 157127, San Francisco, California
  - Duplicate_Cedars-Sinai Medical Center-West Hollywood /ID# 163839, West Hollywood, California
  - Peak Gastroenterology Associates, PC /ID# 165843, Colorado Springs, Colorado
  - Rocky Mountain Pediatric Gastroenterology /ID# 207170, Lone Tree, Colorado
  - Duplicate_Western Connecticut Medical Group /ID# 165879, Danbury, Connecticut
  - Brandon Premier Health Care, PA/Gulf Coast Research Group, LLC /ID# 162262, Brandon, Florida
  - South Lake Pain Institute, Inc /ID# 162808, Clermont, Florida
  - Omega Research Maitland, LLC /ID# 171082, DeBary, Florida
  - Universal Axon Clinical Research /ID# 165428, Doral, Florida
  - Nature Coast Clinical Research - Inverness /ID# 159408, Inverness, Florida
  - SIH Research Mumtaz, Inc /ID# 163083, Kissimmee, Florida
  - Alliance Medical Research /ID# 163837, Lighthouse PT, Florida
  - Cfagi Llc /Id# 202479, Maitland, Florida
  - Sylvester Comprehensive Cancer Center /ID# 155007, Miami, Florida
  - Coral Research Clinic /ID# 158456, Miami, Florida
  - South Florida Research Ph I-IV, Inc. /ID# 161832, Miami, Florida
  - Gastroenterology Group Naples /ID# 165204, Naples, Florida
  - Advanced Research Institute, Inc /ID# 161966, New Port Richey, Florida
  - Endoscopic Research, Inc. /ID# 205906, Orlando, Florida
  - IMIC Inc. Medical Research /ID# 154942, Palmetto Bay, Florida
  - Duplicate_Clinical Research of West Florida, Inc /ID# 208125, Tampa, Florida
  - Clinical Research Of West Florida - Tampa - North Howard Avenue /ID# 205865, Tampa, Florida
  - Atlanta Gastro Assoc /ID# 154724, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 154850, Macon, Georgia
  - Duplicate_Northwestern University /ID# 158261, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 157124, Chicago, Illinois
  - NorthShore University-Endeavor Health Evanston Hospital /ID# 158265, Evanston, Illinois
  - Southwest Gastroenterology /ID# 164781, Oak Lawn, Illinois
  - Cotton O'Neil Clinical Research Center, Digestive Health /ID# 154722, Topeka, Kansas
  - Duplicate_University of Kentucky Chandler Medical Center /ID# 157120, Lexington, Kentucky
  - University of Louisville Hospital /ID# 210525, Louisville, Kentucky
  - GI Alliance /ID# 161963, Baton Rouge, Louisiana
  - Houma Digestive Health Special /ID# 158264, Houma, Louisiana
  - Delricht Research /ID# 206644, New Orleans, Louisiana
  - Nola Research Works, LLC /ID# 161317, New Orleans, Louisiana
  - Louisiana Research Center, LLC /ID# 162237, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group - Chevy Chase /ID# 154832, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 165001, Columbia, Maryland
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 157126, Ann Arbor, Michigan
  - Clin Res Inst of Michigan, LLC /ID# 169179, Chesterfield, Michigan
  - Center for Digestive Health /ID# 154683, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, PLC d.b.a. West Michigan Clinic /ID# 161313, Wyoming, Michigan
  - Mayo Clinic - Rochester /ID# 163086, Rochester, Minnesota
  - St. Louis University /ID# 161883, St Louis, Missouri
  - University of Nebraska Medical Center /ID# 210058, Omaha, Nebraska
  - Vector Clinical Trials /ID# 160170, Las Vegas, Nevada
  - Revival Research Institute, Inc /ID# 210985, Las Vegas, Nevada
  - NY Scientific /ID# 158294, Brooklyn, New York
  - Saratoga Schenectady Gastroenterology Associates - Burnt Hills /ID# 213447, Burnt Hills, New York
  - Intercity Advanced Gastroentertology Center /ID# 215205, Fresh Meadows, New York
  - Duplicate_Northwell Health Division of Gastroenterology at Great Neck /ID# 168738, Great Neck, New York
  - NYU Langone Long Island Clinical Research Associates /ID# 154829, Lake Success, New York
  - Digestive Disease Care /ID# 211777, New Hyde Park, New York
  - NYU Langone Medical Center /ID# 160169, New York, New York
  - Weill Cornell Medicine /ID# 165878, New York, New York
  - Icahn School of Medicine at Mount Sinai /ID# 165612, New York, New York
  - Columbia Univ Medical Center /ID# 161899, New York, New York
  - Lenox Hill Hospital /ID# 168467, New York, New York
  - Duplicate_DiGiovanna Institute for Medical Education & Research /ID# 171126, North Massapequa, New York
  - Univ NC Chapel Hill /ID# 154833, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 158428, Charlotte, North Carolina
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 154873, Raleigh, North Carolina
  - Plains Clinical Research Center, LLC /ID# 169718, Fargo, North Dakota
  - Tri-State Endoscopy Center /ID# 154927, Cincinnati, Ohio
  - Cleveland Clinic Main Campus /ID# 209226, Cleveland, Ohio
  - The Ohio State University /ID# 164708, Columbus, Ohio
  - Optimed Research, Ltd. /ID# 167887, Columbus, Ohio
  - Hometown Urgent Care and Resea /ID# 170464, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC /ID# 201770, Mentor, Ohio
  - Hightower Clinical /ID# 211993, Oklahoma City, Oklahoma
  - Digestive Disease Specialists /ID# 170775, Oklahoma City, Oklahoma
  - Adult Gastroenterology Associates - Gen 1 Research /ID# 208864, Tulsa, Oklahoma
  - Children's Hospital of Pittsburgh of UPMC /ID# 212544, Pittsburgh, Pennsylvania
  - Digestive Disease Associates, LTD - Wyomissing /ID# 208297, Wyomissing, Pennsylvania
  - Medical University of South Carolina /ID# 212858, Charleston, South Carolina
  - Gastroenterology Associates, P.A. of Greenville /ID# 154904, Greenville, South Carolina
  - Rapid City Medical Center - GI Research /ID# 163838, Rapid City, South Dakota
  - Gastro One /ID# 154726, Cordova, Tennessee
  - East Tennessee Research Institute /ID# 168739, Johnson City, Tennessee
  - Clinical Neuroscience Solutions - Memphis /ID# 164180, Memphis, Tennessee
  - Vanderbilt University Medical Center /ID# 157121, Nashville, Tennessee
  - TX Clinical Research Institute /ID# 159404, Arlington, Texas
  - Inquest Clinical Research /ID# 165694, Baytown, Texas
  - Texas Digestive Disease Consultants /ID# 209946, Cedar Park, Texas
  - GI Alliance /ID# 209797, Cedar Park, Texas
  - Baylor Scott & White Center for Inflammatory Bowel Diseases /ID# 159406, Dallas, Texas
  - Duplicate_DHAT Research Institute /ID# 158208, Garland, Texas
  - Vilo Research Group Inc /ID# 207655, Houston, Texas
  - Baylor College of Medicine /ID# 158203, Houston, Texas
  - Centex Studies, Inc. - Houston /ID# 201219, Houston, Texas
  - Clinical Associates in Research Therapeutics of America, LLC /ID# 161323, San Antonio, Texas
  - Southern Star Research Institute, LLC /ID# 168773, San Antonio, Texas
  - Baylor Scott & White Center for Diagnostic Medicine /ID# 204131, Temple, Texas
  - Tyler Research Institute, LLC /ID# 166797, Tyler, Texas
  - Gastro Health & Nutrition - Victoria /ID# 164290, Victoria, Texas
  - Advanced Research Institute /ID# 154907, Ogden, Utah
  - Velocity Clinical Research - Salt Lake City /ID# 161778, West Jordan, Utah
  - Richmond VA Medical Center /ID# 159988, Richmond, Virginia
  - Duplicate_Virginia Mason Medical Center /ID# 155556, Seattle, Washington
  - West Virginia University Hospitals /ID# 167941, Morgantown, West Virginia
- Argentina (4):
  - Cemic /Id# 168078, Ciudad Autonoma Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires /ID# 168077, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Hospital Provincial del Centenario /ID# 170886, Rosario, Santa Fe Province
  - Hospital Privado Universitario - Hospital Privado Centro Medico de Cordoba S.A. /ID# 168076, Córdoba
- Australia (4):
  - Mater Misericordiae Limited /ID# 167220, South Brisbane, Queensland
  - Griffith University /ID# 212635, Southport, Queensland
  - Lyell McEwin Hospital /ID# 212215, Elizabeth Vale, South Australia
  - Emeritus Research /ID# 213512, Camberwell, Victoria
- Austria (4):
  - Universitaetsklinikum St. Poelten /ID# 166424, Sankt Pölten, Lower Austria
  - Medizinische Universitaet Graz /ID# 158140, Graz, Styria
  - Krankenhaus der Barmherzigen Brueder Wien /ID# 212060, Vienna, Vienna
  - Medizinische Universitaet Wien /ID# 158141, Vienna, Vienna
- Belarus (3):
  - Grodno city clinical hospital #2 /ID# 205113, Hrodna, Grodnenskaya
  - Gomel Regional Clinical Hospital /ID# 205112, Homyel
  - Vitebsk Regional Advanced Clin /ID# 206778, Vitebsk
- Belgium (13):
  - Imelda Ziekenhuis /ID# 157403, Bonheiden, Antwerpen
  - AZ Sint-Maarten /ID# 212876, Mechelen, Antwerpen
  - ZAS Palfijn /ID# 212877, Merksem, Antwerpen
  - Universite Libre de Bruxelles - Hopital Erasme /ID# 157408, Anderlecht, Brussels Capital
  - Cliniques Universitaires UCL Saint-Luc /ID# 157406, Brussels, Brussels Capital
  - Groupe Sante CHC - Clinique du MontLegia /ID# 157404, Liège, Liege
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant /ID# 157412, Yvoir, Namur
  - UZ Gent /ID# 157405, Ghent, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 157407, Leuven, Vlaams-Brabant
  - AZ-Delta /ID# 157402, Roeselare, West-Vlaanderen
  - AZ Maria Middelares /ID# 213532, Ghent
  - AZ Groeninge /ID# 211513, Kortrijk
  - CHU de Liege /ID# 157409, Liège
- Bosnia and Herzegovina (2):
  - Klinicki centar Banja Luka /ID# 164513, Banja Luka, Republika Srpska
  - Clinical Center University of Sarajevo /ID# 165139, Sarajevo
- Bulgaria (7):
  - UMHAT Dr Georgi Stranski EAD /ID# 203976, Pleven
  - Umbal Kaspela /ID# 165700, Plovdiv
  - 2nd Mhat /ID# 165702, Sofia
  - Tokuda Hospital Sofia /ID# 165701, Sofia
  - UMHAT Sveti Ivan Rilski /ID# 204815, Sofia
  - Duplicate_UMHAT Tsaritsa Joanna - ISUL /ID# 211242, Sofia
  - MHAT Trakia /ID# 201668, Stara Zagora
- Canada (19):
  - University of Calgary /ID# 157155, Calgary, Alberta
  - Allen Whey Khye Lim Professional Corporation /ID# 169763, Edmonton, Alberta
  - University of Alberta Hospital /ID# 157099, Edmonton, Alberta
  - Covenant Health /ID# 161632, Edmonton, Alberta
  - Fraser Clinical Trials Inc /ID# 159055, New Westminster, British Columbia
  - Giri Gi Research Institute - Vancouver /ID# 157096, Vancouver, British Columbia
  - Percuro Clinical Research, Ltd /ID# 161631, Victoria, British Columbia
  - Queen Elizabeth II Health Sciences Centre - Victoria General /ID# 157088, Halifax, Nova Scotia
  - IWK Health Center /ID# 165905, Halifax, Nova Scotia
  - Medicor Research Inc /ID# 157150, Greater Sudbury, Ontario
  - Duplicate_Hamilton Health Sciences -McMaster University Medical Centre /ID# 157184, Hamilton, Ontario
  - London Health Sciences Center- University Hospital /ID# 157161, London, Ontario
  - Scott Shulman Medicine Professional Corporation /ID# 165906, North Bay, Ontario
  - Mount Sinai Hospital /ID# 169764, Toronto, Ontario
  - Toronto Digestive Disease Associates /ID# 157158, Vaughan, Ontario
  - Hotel Dieu de Levis /ID# 214377, Lévis, Quebec
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 159056, Montreal, Quebec
  - Montreal General Hospital- McGill University Health Center /ID# 157085, Montreal, Quebec
  - CISSS de la Monteregie Centre - Hopital Charles Le Moyne /ID# 161630, Greenfield Park
- Chile (4):
  - Hospital Guillermo Grant Benavente de Concepción /ID# 210760, Concepción, Bio-Bio
  - Hospital Las Higueras /ID# 167092, Talcahuano, Bio-Bio
  - Servicio de Salud Occidente Hospital San Juan de Dios /ID# 171122, Santiago, Region Metropolitana Santiago
  - Complejo Asistencial Dr. Sotero del Rio /ID# 169384, Santiago, Santiago Metropolitan
- China (16):
  - Guangdong Provincial People's Hospital /ID# 212949, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University /ID# 210784, Guangzhou, Guangdong
  - The Second Hospital of Hebei Medical University /ID# 212738, Shijiazhuang, Hebei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 211039, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 210858, Wuhan, Hubei
  - Renmin Hospital of Wuhan University /ID# 214874, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University /ID# 211700, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University /ID# 211036, Nanchang, Jiangxi
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine /ID# 210840, Shanghai, Shanghai Municipality
  - Renji Hospital, Shanghai Jiaotong University School of Medicine /ID# 210705, Shanghai, Shanghai Municipality
  - Shanghai East Hospital /ID# 212684, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University /ID# 210890, Chengdu, Sichuan
  - Tianjin Medical University General Hospital /ID# 210926, Tianjin, Tianjin Municipality
  - The second affiliated hospital of Zhejiang University school of medicine /ID# 210724, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine /ID# 210625, Hangzhou, Zhejiang
  - Jinhua Municipal Central Hospital /ID# 215628, Jinhua, Zhejiang
- Colombia (4):
  - Instituto de Coloproctologia /ID# 158743, Medellín, Antioquia
  - Hospital Pablo Tobón Uribe /ID# 158730, Medellín, Antioquia
  - Hospital Universitario San Vic /ID# 171486, Medellín, Antioquia
  - Hospital Univ San Ignacio /ID# 158734, Bogota, Cundinamarca
- Croatia (6):
  - Klinicka bolnica Dubrava Zagreb /ID# 157560, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre milosrdnice /ID# 157728, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb /ID# 157561, Zagreb, City of Zagreb
  - Poliklinika Borzan d.o.o. /ID# 157559, Osijek, County of Osijek-Baranja
  - Klinicki Bolnicki Centar (KBC) Split /ID# 157562, Split, Split-Dalmatia County
  - Zadar General Hospital /ID# 157563, Zadar
- Czechia (9):
  - Duplicate_Institut klinicke a experimentalni mediciny (IKEM) /ID# 165465, Prague, Praha 4
  - Iscare Klinické Centrum /ID# 225794, Prague, Praha 9
  - Hepato-Gastroenterologie HK, s.r.o. /ID# 163225, Hradec Králové
  - Nemocnice Pardubickeho kraje, a.s. /ID# 163226, Pardubice
  - Nemocnice Milosrdnych sester sv. Karla Boromejskeho v Praze /ID# 211306, Prague
  - Axon Clinical, s.r.o. /ID# 163223, Prague
  - Fakultni Thomayerova nemocnice /ID# 162941, Prague
  - ResTrial s.r.o. /ID# 211078, Prague
  - Nemocnice Horovice - NH Hospital a.s /ID# 211077, Prague
- Denmark (5):
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 155530, Hvidovre, Capital Region
  - Aarhus Universitetshospital - Skejby /ID# 155664, Aarhus, Central Jutland
  - Roskilde Sygehus /ID# 155532, Roskilde, Region Sjælland
  - Sygehusenheden Nyborg - OUH /ID# 161525, Nyborg, Region Syddanmark
  - Odense University Hospital /ID# 155531, Odense, Region Syddanmark
- Egypt (6):
  - Alexandria University /ID# 157187, Alexandria, Alexandria Governorate
  - Alexandria University /ID# 164540, Alexandria, Alexandria Governorate
  - Zagazig University Hospitals /ID# 164539, Al Sharqia
  - Clinical Research Center, Faculty of Medicine, Cairo university /ID# 157175, Cairo
  - National Hepatology and Tropical Medicine Research Institute /ID# 157874, Cairo
  - Duplicate_Internal Medicine Department, Faculty of Medicine, AinShams University /ID# 157506, Cairo
- Estonia (3):
  - North Estonia Medical Centre /ID# 164326, Mustamäe, Harju
  - West Tallinn Central Hospital /ID# 157075, Tallinn, Harju
  - East Tallinn Central Hospital /ID# 157074, Tallinn
- France (12):
  - Chu de Nice-Hopital L'Archet Ii /Id# 162557, Nice, Alpes-Maritimes
  - Centre Hospitalier Universitaire de Bordeaux /ID# 162558, Pessac, Gironde
  - CHU Montpellier - Hopital Saint Eloi /ID# 215147, Montpellier, Herault
  - Duplicate_CHU Grenoble - Hopital Michallon /ID# 212834, La Tronche, Isere
  - CHRU Nancy - Hopitaux de Brabois /ID# 162561, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 162559, Lille, Nord
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 162562, St-Priest-en-Jarez, Pays de la Loire Region
  - HCL - Hopital Lyon Sud /ID# 162560, Pierre-Bénite, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 165058, Amiens, Somme
  - CHRU Pontchaillou /ID# 213209, Rennes
  - Hopital Beaujon /ID# 166284, Clichy, Île-de-France Region
  - Centre Medico Chirurgical Ambroise Pare Hartmann /ID# 249858, Neuilly-sur-Seine, Île-de-France Region
- Germany (28):
  - Universitaetsklinikum Freiburg /ID# 162030, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis fuer Gastroenterologie /ID# 166150, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 162031, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 164990, Ulm, Baden-Wurttemberg
  - Medizinisches Versorgunszentrum Dachau /ID# 211555, Dachau, Bavaria
  - Universitaetsklinikum Erlangen /ID# 159343, Erlangen, Bavaria
  - Duplicate_Agaplesion Markus Krankenhaus /ID# 159345, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt /ID# 212979, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover /ID# 162032, Hanover, Lower Saxony
  - Klinikum Lueneburg /ID# 163678, Lüneburg, Lower Saxony
  - Universitaetsklinikum Koeln /ID# 164989, Cologne, North Rhine-Westphalia
  - Evangelisches Krankenhaus Kalk /ID# 212726, Cologne, North Rhine-Westphalia
  - Praxiszentrum fuer Gastroenterologie /ID# 211966, Grevenbroich, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 162029, Minden, North Rhine-Westphalia
  - Universitaetsklinikum Muenster /ID# 159344, Münster, North Rhine-Westphalia
  - Zentrum für Gastroenterologie Saar MVZ GmbH /ID# 210528, Saarbrücken, Saarland
  - Eugastro /ID# 212078, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel /ID# 159349, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 159351, Jena, Thuringia
  - Duplicate_Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 212220, Berlin
  - Duplicate_Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 212894, Berlin
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 211974, Berlin
  - MVZ fuer Gastroenterlogie am Bayerischen Platz /ID# 159350, Berlin
  - DRK Kliniken Berlin Westend /ID# 166151, Berlin
  - Krankenhaus Waldfriede /ID# 212727, Berlin-Zehlendorf
  - Stadtisches Klinikum Braunschweig /ID# 163680, Braunschweig
  - Universitaetsklinikum Magdeburg /ID# 211843, Magdeburg
  - Universitaetsklinikum Regensburg /ID# 163813, Regensburg
- Greece (7):
  - General Hospital of Chest Diseases of Athens SOTIRIA /ID# 170914, Athens, Attica
  - General Hospital of Nikaia-Piraeus "Agios Panteleimon" /ID# 157424, Nikaia, Attica
  - Tzaneio general hospital of Piraeus /ID# 206443, Piraeus, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 157422, Heraklion, Crete
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 157423, Athens
  - University General Hospital of Ioannina /ID# 157420, Ioannina
  - Theageneio Anticancer Hospital /ID# 163897, Thessaloniki
- Hong Kong (2):
  - Queen Mary Hospital /ID# 163923, Hong Kong
  - Tuen Mun Hospital /ID# 163905, Hong Kong
- Ireland (3):
  - Duplicate_Beaumont Hospital /ID# 157543, Beaumont, Dublin
  - St Vincent's University Hospital /ID# 157540, Elm Park, Dublin
  - University Hospital Galway /ID# 157541, Galway
- Israel (9):
  - Shaare Zedek Medical Center /ID# 163541, Jerusalem, Jerusalem
  - Shaare Zedek Medical Center /ID# 171068, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 165914, Jerusalem, Jerusalem
  - The Edith Wolfson Medical Center /ID# 217331, Ashkelon, Southern District
  - Soroka University Medical Center /ID# 157794, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 157793, Ramat Gan, Tel Aviv
  - The Chaim Sheba Medical Center /ID# 171069, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 157792, Tel Aviv, Tel Aviv
  - Duplicate_Rambam Medical Center /ID# 171067, Haifa
- Italy (19):
  - Duplicate_AOU Ospendali Riuniti di Ancona /ID# 162436, Torrette, Ancona
  - Duplicate_Ospedale Policlinico San Martino /ID# 162439, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 155642, Rozzano, Lombardy
  - ASST Fatebenefratelli Sacco /ID# 155639, Milan, Milano
  - ASST Rhodense/Presidio Ospedaliero di Rho /ID# 212227, Rho, Milano
  - Duplicate_Fondazione Policlinico Universitario Campus Bio-Medico di Roma /ID# 162438, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 158022, Rome, Roma
  - Azienda Ospedaliera San Camillo Forlanini /ID# 155644, Rome, Roma
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 166912, Rome, Roma
  - Presidio Columbus-Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Un /ID# 155640, Rome, Roma
  - Duplicate_Azienda Ospedaliera Univ. Meyer /ID# 167992, Florence, Tuscany
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 161299, Negrar, Verona
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 155643, Bologna
  - Ospedale Cannizzaro /ID# 161300, Catania
  - Azienda Ospedaliero-Universitaria Renato Dulbecco /ID# 212016, Catanzaro
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 155641, Milan
  - Duplicate_Azienda Ospedaliero-Universitaria Policlinico di Modena /ID# 212028, Modena
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 155645, Palermo
  - Duplicate_Fondazione IRCCS Policlinico S. Matteo /ID# 212031, Pavia
- Japan (45):
  - Aichi Medical University Hospital /ID# 160097, Nagakute, Aichi-ken
  - Daido Clinic - Nagoya /ID# 211476, Nagoya, Aichi-ken
  - Nagoya University Hospital /ID# 160116, Nagoya, Aichi-ken
  - Nagoya City University Hospital /ID# 160100, Nagoya, Aichi-ken
  - Duplicate_Fujita Health University Hospital /ID# 163234, Toyoake-shi, Aichi-ken
  - Tokatsu Tsujinaka Hospital /ID# 163352, Abiko-shi, Chiba
  - Duplicate_Chiba University Hospital /ID# 217533, Chiba, Chiba
  - Tsujinaka Hospital - Kashiwanoha /ID# 213848, Kashiwa-shi, Chiba
  - The Jikei University Kashiwa Hospital /ID# 200030, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 160099, Sakura-shi, Chiba
  - Fukuoka University Hospital /ID# 217793, Fukuoka, Fukuoka
  - Kurume University Hospital /ID# 160106, Kurume-shi, Fukuoka
  - National Hospital Organization Fukuyama Medical Center /ID# 163577, Fukuyama-shi, Hiroshima
  - Hiroshima University Hospital /ID# 160109, Hiroshima, Hiroshima
  - Duplicate_Asahikawa Medical University Hospital /ID# 162848, Asahikawa-shi, Hokkaido
  - Sapporo Tokushukai Hospital /ID# 213492, Sapporo, Hokkaido
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital /ID# 160096, Sapporo, Hokkaido
  - Sapporo Medical University Hospital /ID# 163056, Sapporo, Hokkaido
  - Nishinomiya Municipal Central Hospital /ID# 210103, Nishinomiya-shi, Hyōgo
  - Hyogo Medical University Hospital /ID# 160107, Nishinomiya-shi, Hyōgo
  - NHO Mito Medical Center /ID# 160092, Higashiibaraki-gun, Ibaraki
  - Kanazawa University Hospital /ID# 202258, Kanazawa, Ishikawa-ken
  - Gokeikai Ofuna Chuo Hospital /ID# 171066, Kamakura-shi, Kanagawa
  - Kitasato University Hospital /ID# 171065, Sagamihara-shi, Kanagawa
  - Duplicate_Yokohama Municipal Citizen's Hospital /ID# 207161, Yokohama, Kanagawa
  - Duplicate_Yokohama City University Medical Center /ID# 163907, Yokohama, Kanagawa
  - Mie University Hospital /ID# 203640, Tsu, Mie-ken
  - Yokkaichi Hazu Medical Center /ID# 163764, Yokkaichi-shi, Mie-ken
  - Tohoku University Hospital /ID# 162847, Sendai, Miyagi
  - Tohoku Rosai Hospital /ID# 163229, Sendai, Miyagi
  - Osaka Metropolitan University Hospital /ID# 160117, Osaka, Osaka
  - Saitama Medical Center /ID# 160093, Kawagoe, Saitama
  - Tokitokai Tokito clinic /ID# 160110, Saitama-shi, Saitama
  - Shiga University of Medical Science Hospital /ID# 164025, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 205690, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 163057, Sunto-gun, Shizuoka
  - Institute of Science Tokyo Hospital /ID# 160095, Bunkyo-ku, Tokyo
  - Tokai University Hachioji Hospital /ID# 160098, Hachioji-shi, Tokyo
  - The Jikei University Hospital /ID# 163209, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 160105, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 160114, Mitaka-shi, Tokyo
  - Tokyo Women's Medical University Hospital /ID# 205974, Shinjuku-ku, Tokyo
  - Wakayama Medical University Hospital /ID# 202561, Wakayama, Wakayama
  - Yamagata University Hospital /ID# 200159, Yamagata, Yamagata
  - Yamanashi Prefectural Central Hospital /ID# 160094, Kofu, Yamanashi
- Latvia (3):
  - VCA Polyclinic Aura /ID# 159611, Riga
  - Pauls Stradins Clinical University Hospital /ID# 159612, Riga
  - Duplicate_Digestive Disease Center Gastro /ID# 163107, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics /ID# 162583, Kaunas
  - Vilnius University Hospital Santaros Klinikos /ID# 162514, Vilnius
- Malaysia (3):
  - Universiti Sains Malaysia /ID# 160666, Kelantan, Kelantan
  - Queen Elizabeth Hospital /ID# 160664, Division Pantai Barat Utara, Sabah
  - Universiti Kebangsaan Malaysia (UKM) Medical Centre /ID# 201363, Kuala Lumpur, Selangor
- Mexico (4):
  - Investigacion Biomedica para el Desarrollo de Farmacos, S.A. de C.V. /ID# 170734, Zapopan, Jalisco
  - JM Research SC /ID# 170729, Cuernavaca, Morelos
  - Unidad de Atencion Medica e Investigacion en Salud /ID# 170732, Mérida, Yucatán
  - Health Pharma Professional Research S.A de C.V /ID# 170730, Del. Benito Juárez
- Netherlands (2):
  - Elisabeth Tweesteden Ziekenhuis /ID# 163632, Tilburg, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 157956, Amsterdam, North Holland
- New Zealand (4):
  - Aotearoa Clinical Trials /ID# 167226, Papatoetoe, Auckland
  - Christchurch Hospital. /ID# 167224, Christchurch, Canterbury
  - Dunedin Hospital /ID# 167227, Otago, Otago
  - Duplicate_Wellington Hospital (Capital and Coast District Health Board) /ID# 167225, Wellington
- Norway (4):
  - Duplicate_Vestre viken - Baerum Sykehus /ID# 212996, Gjettum, Akershus
  - Akershus Universitetssykehus /ID# 169379, Nordbyhagen, Akershus
  - Helse More og Romsdal HF, Alesund sjukehus /ID# 212810, Ålesund, Møre og Romsdal
  - Sykehuset Levanger Helse NT /ID# 201669, Levanger, Nord-Trondelag
- Poland (15):
  - Solumed Centrum Medyczne /ID# 163569, Poznan, Greater Poland Voivodeship
  - Gastromed Sp. z o.o /ID# 212476, Torun, Kuyavian-Pomeranian Voivodeship
  - Duplicate_Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wrocl /ID# 212601, Wroclaw, Lower Silesian Voivodeship
  - Planetmed Sp. z o.o. /ID# 202799, Wroclaw, Lower Silesian Voivodeship
  - 1 Wojskowy Szpital Kliniczny Z Poliklinika /Id# 210940, Lublin, Lublin Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 4 W Lublinie /ID# 210941, Lublin, Lublin Voivodeship
  - Centrum Zdrowia MDM /ID# 163570, Warsaw, Masovian Voivodeship
  - Panstwowy Instytut Medyczny MSWiA w Warszawie /ID# 163582, Warsaw, Masovian Voivodeship
  - Vivamed Sp. z o.o. /ID# 202800, Warsaw, Masovian Voivodeship
  - Instytut Pomnik - Centrum Zdrowia Dziecka /ID# 213580, Warsaw, Masovian Voivodeship
  - Centrum Medycznym Medyk /ID# 212891, Rzeszów, Podkarpackie Voivodeship
  - Centrum Medyczne Lukamed Sp. z o.o. /ID# 212478, Chojnice, Pomeranian Voivodeship
  - H-T Centrum Medyczne Endoterapia /ID# 212475, Tychy, Silesian Voivodeship
  - Wojewódzki Szpital Specjalistyczny W Olsztynie /ID# 212474, Olsztyn, Warmian-Masurian Voivodeship
  - Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego w Lodzi /ID# 212477, Lodz, Łódź Voivodeship
- Portugal (11):
  - Duplicate_Hospital da Senhora da Oliveira Guimaraes, EPE /ID# 160737, Guimarães, Braga District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital de Portimão /ID# 167752, Portimão, Faro District
  - Centro Hospitalar de Entre Douro e Vouga /ID# 160672, Santa Maria DA Feira, Porto District
  - Duplicate_Hospital Garcia de Orta, EPE /ID# 160745, Almada, Setúbal District
  - Centro Hospitalar Universitário do Algarve, EPE - Hospital Faro /ID# 160713, Faro
  - Centro Hospitalar de Lisboa Central /ID# 160673, Lisbon
  - Centro Hospitalar de Lisboa Ocidental, EPE - Hospital Egas Moniz /ID# 167751, Lisbon
  - Unidade Local de Saude de Santa Maria, EPE /ID# 160692, Lisbon
  - Hospital de Loures, E.P.E /ID# 207759, Loures
  - Unidade Local de Saude Sao Joao, EPE /ID# 160693, Porto
  - Centro Hosp de Tondela-Viseu /ID# 160699, Viseu
- Romania (4):
  - Fundeni Clinical Institute /ID# 170899, Bucharest
  - Tvm Med Serv Srl /Id# 170902, Cluj-Napoca
  - Cabinet Particular Policlinic Algomed /ID# 170900, Timișoara
  - Duplicate_Centrul Medical Tuculanu SRL /ID# 170903, Timișoara
- Russia (11):
  - Kuzbass Regional Clinical Hospital /ID# 200962, Kemerovo, Kemerovo Oblast
  - Novosibirski Gastrocenter /ID# 217552, Novosibirsk, Novosibirsk Oblast
  - Duplicate_Perm state medical university n.a. E.A. Vagner /ID# 207439, Perm, Permskiy Kray
  - Duplicate_St. Petersburg State Pediatric Medical University /ID# 211978, Saint Petersburg, Sankt-Peterburg
  - Professor Pasechnikov Gastroenterology and Pankreatology clinic /ID# 200970, Stavropol, Stavropol Kray
  - Tver Regional Clinical Hospital /ID# 206858, Tver', Tver Oblast
  - Regional Clinical Hospital #1 /ID# 200973, Tyumen, Tyumen Oblast
  - Alliance Biomedical Ural Group /ID# 200972, Izhevsk, Udmurtiya Republic
  - National Medical Research Center of Coloproctology n.a. A. N. Ryzhikh /ID# 204808, Moscow
  - City Clinical Hospital No. 31 /ID# 208872, Saint Petersburg
  - Ulyanovsk Regional Clinical Hospital /ID# 200964, Ulyanovsk
- Serbia (9):
  - Clinical Hosp Center Zvezdara /ID# 157052, Belgrade, Beograd
  - Military Medical Academy /ID# 157053, Belgrade, Beograd
  - University Children's Hospital 'Tirsova' /ID# 211482, Belgrade, Beograd
  - University Clinical Center Serbia /ID# 157047, Belgrade, Beograd
  - Clinical Hospital Center Dr Dragisa Misovic - Dedinje /ID# 212799, Belgrade, Beograd
  - Clin Hosp Ctr Bezanijska Kosa /ID# 157050, Belgrade, Beograd
  - General Hospital Leskovac /ID# 209575, Leskovac, Jablanicki Okrug
  - Duplicate_University Clinical Center Kragujevac /ID# 157049, Kragujevac, Sumadijski Okrug
  - University Clinical Center Vojvodina /ID# 157046, Novi Sad
- Singapore (3):
  - Mount Elizabeth Hospital /ID# 205741, Singapore, Central Singapore
  - National University Hospital /ID# 160667, Singapore
  - Singapore General Hospital /ID# 160668, Singapore
- Slovakia (3):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica /ID# 156468, Banská Bystrica, Banská Bystrica Region
  - KM Management, spol. s.r.o. /ID# 206764, Nitra, Nitra Region
  - Gastro I., s.r.o. /ID# 156469, Prešov, Presov
- South Africa (4):
  - Clinresco Centers /ID# 163865, Johannesburg, Gauteng
  - Wits Clinical Research /ID# 158114, Johannesburg, Gauteng
  - Private Practice Dr MN Rajabally /ID# 163112, Cape Town, Western Cape
  - Spoke Research Inc /ID# 158116, CAPE TOWN Milnerton, Western Cape
- South Korea (12):
  - Inje University Haeundae Hospital /ID# 202518, Busan, Busan Gwang Yeogsi
  - Dong-A University Medical Center /ID# 158699, Busan, Busan Gwang Yeogsi
  - Pusan National University Hospital /ID# 158695, Busan, Busan Gwang Yeogsi
  - The Catholic University of Korea, Daejeon St. Mary's Hospital /ID# 213554, Daejeon, Daejeon Gwang Yeogsi
  - Hanyang University Guri Hospital /ID# 158690, Guri-si, Gyeonggido
  - Duplicate_CHA University Bundang Medical Center /ID# 158698, Seongnam-si, Gyeonggido
  - The Catholic University Of Korea St. Vincent's Hospital /ID# 158693, Suwon, Gyeonggido
  - Kangbuk Samsung Hospital /ID# 158694, Seoul, Seoul Teugbyeolsi
  - Asan Medical Center /ID# 158696, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 158692, Seoul, Seoul Teugbyeolsi
  - Yeungnam University Medical Center /ID# 158691, Daegu
  - Yonsei University Health System Severance Hospital /ID# 158689, Seoul
- Spain (14):
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 157553, Ferrol, A Coruna
  - Hospital Universitari de Bellvitge /ID# 208207, L'Hospitalet de Llobregat, Barcelona
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 159237, Sabadell, Barcelona
  - Hospital Universitario Puerta de Hierro - Majadahonda /ID# 157573, Majadahonda, Madrid
  - Hospital Universitario Basurto /ID# 205190, Bilbao, Vizcaya
  - Hospital Clinic de Barcelona /ID# 157552, Barcelona
  - Hospital General Universitario Gregorio Maranon /ID# 161145, Madrid
  - Hospital Universitario La Paz /ID# 159235, Madrid
  - Hospital Universitario de Salamanca /ID# 157558, Salamanca
  - Hospital Universitario Virgen Macarena /ID# 159967, Seville
  - Hospital Clinico Universitario de Valencia /ID# 209700, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 157556, Valencia
  - Hospital Clinico Universitario Lozano Blesa /ID# 212525, Zaragoza
  - Hospital Universitario Miguel Servet /ID# 157557, Zaragoza
- Sweden (7):
  - Skane University hospital /ID# 211745, Malmo, Skåne County
  - Karolinska University Hospital Solna /ID# 212025, Solna, Stockholm County
  - GHP Stockholm Gastro Center /ID# 211748, Stockholm, Stockholm County
  - Medicinkliniken, Gastroenheten /ID# 163744, Stockholm, Stockholm County
  - Danderyd Hospital /ID# 202138, Stockholm, Stockholm County
  - Duplicate_Sahlgrenska University Hospital /ID# 163792, Gothenburg, Västra Götaland County
  - Duplicate_Sahlgrenska University Hospital /ID# 163797, Gothenburg, Västra Götaland County
- Switzerland (3):
  - University Hospital Basel /ID# 164554, Basel Town, Canton of Basel-City
  - University Hospital Zurich /ID# 163536, Zurich, Canton of Zurich
  - Inselspital, Universitaetsspital Bern /ID# 163535, Bern
- Taiwan (5):
  - National Taiwan University Hospital /ID# 162190, Taipei City, Taipei
  - China Medical University Hospital /ID# 160141, Taichung
  - Taichung Veterans General Hospital /ID# 160140, Taichung
  - National Cheng Kung University Hospital /ID# 160142, Tainan
  - Taipei Veterans General Hosp /ID# 212712, Taipei
- Ukraine (12):
  - Lviv Railway Clinical Hospital of branch Healthcare Centers of Public Joint Stoc /ID# 165658, Lviv, Lviv Oblast
  - MNE Vinnytsia Regional Clinical Hospital n.a. M.I.Pyrogov /ID# 216474, Vinnytsia, Vinnytsia Oblast
  - University Hospital of M.I. Pyrogov VNMU /ID# 212000, Vinnytsia, Vinnytsia Oblast
  - ME Volyn Regional Clinical Hospital of Volyn Regional Council /ID# 206789, Lutsk, Volyn Oblast
  - Transcarpathian Regional Clinical Hospital n.a. Andriy Novak /ID# 167960, Uzhhorod, Zakarpattia Oblast
  - Kharkiv City Clinical Hospital No.2 n.a. Prof. O.O. Shalimov /ID# 165657, Kharkiv
  - Municipal Nonprofit Enterprise Kherson city clinical hospital n.a. Y.Y. Karabel /ID# 212399, Kherson
  - Kyiv City Clinical Hospital No.18 /ID# 162531, Kyiv
  - Medical Center OK Clinic LLC, International Institute of Clinical Research /ID# 211998, Kyiv
  - Communal Noncommercial Institution Consultative and Diagnostic Center of Desnian /ID# 165659, Kyiv
  - Medical Center of LLC Medbud-Clinic /ID# 216998, Kyiv
  - Kyiv Railway Clinical Hosp No.2 /ID# 217366, Kyiv
- United Kingdom (16):
  - Addenbrooke's Hospital /ID# 158034, Cambridge, Cambridgeshire
  - Duplicate_Royal Devon University Healthcare NHS Foundation Trust /ID# 157544, Exeter, Devon
  - Hull University Teaching Hospitals NHS Trust /ID# 158761, Hull, East Riding Of Yorkshire
  - Western General Hospital - NHS Lothian /ID# 207448, Edinburgh, Edinburgh, City of
  - Gartnavel General Hospital /ID# 202568, Glasgow, Glasgow City
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 163713, London, Greater London
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 157546, London, Greater London
  - Oxford University Hospitals NHS Foundation Trust /ID# 158036, Oxford, Oxfordshire
  - Ashford and St Peter's Hospitals NHS Foundation Trust /ID# 207936, Chertsey, Surrey
  - Leeds Teaching Hospitals NHS Trust /ID# 157550, Leeds, West Yorkshire
  - Barnsley Hospital NHS Foundation Trust /ID# 202773, Barnsley
  - University Hospitals Birmingham NHS Foundation Trust /ID# 157545, Birmingham
  - Calderdale and Huddersfield NHS Foundation Trust /ID# 209570, Huddersfield
  - King's College Hospital NHS Foundation Trust /ID# 158760, London
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust /ID# 163708, Newcastle upon Tyne
  - Northern Care Alliance NHS Group /ID# 207766, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Panaccione R, Ferrante M, Dotan I, Panes J, Hisamatsu T, Bossuyt P, Danese S, Song A, Kalabic J, Joshi N, Zambrano J, Zhang Y, Duan WR, Kligys K, Dubinsky MC, Lindsay JO, Vermeire S, Siegmund B, Irving PM, D'Haens G. Extended Risankizumab Treatment in Patients With Crohn's Disease Who Did Not Achieve Clinical Response to Induction Treatment. Clin Gastroenterol Hepatol. 2025 Oct;23(11):2012-2022.e6. doi: 10.1016/j.cgh.2024.12.023. Epub 2025 Feb 3. PMID 39909280
- [Derived] Feagan BG, Colombel JF, Panaccione R, Schreiber S, Ferrante M, Kamikozuru K, Ma C, Lee WJ, Griffith J, Joshi N, Kligys K, Kalabic J, Xuan S, Dubinsky M. Early Endoscopic Outcomes After Risankizumab Are Associated With Fewer Hospitalizations and Surgeries in Crohn's Disease. Gastro Hep Adv. 2024 Sep 5;4(1):100544. doi: 10.1016/j.gastha.2024.08.022. eCollection 2025. PMID 39802486
- [Derived] Atreya R, Ferrante M, Panaccione R, Feagan B, Shchukina O, Jairath V, Rieder F, Hisamatsu T, Siegmund B, Kligys K, Song A, Zambrano J, Mallick M, Zhang Y, Armuzzi A, D'Haens G. Risankizumab Is Associated With Normalization of Biomarkers in Patients With Crohn's Disease: Results From the Phase 3 ADVANCE, MOTIVATE, and FORTIFY Studies. J Crohns Colitis. 2025 Apr 4;19(4):jjae164. doi: 10.1093/ecco-jcc/jjae164. PMID 39485390
- [Derived] Peyrin-Biroulet L, Colombel JF, Louis E, Ferrante M, Motoya S, Panaccione R, Torres J, Ungaro RC, Kligys K, Kalabic J, Zambrano J, Zhang Y, D'Haens G. Shorter Crohn's Disease Duration Is Associated With Better Clinical and Endoscopic Outcomes With Risankizumab in Phase 3 Studies. Gastro Hep Adv. 2024 Mar 7;3(4):539-550. doi: 10.1016/j.gastha.2024.02.008. eCollection 2024. PMID 39131711
- [Derived] Ferrante M, Irving PM, Abreu MT, Axler J, Gao X, Cao Q, Fujii T, Rausch A, Torres J, Neimark E, Song A, Wallace K, Kligys K, Berg S, Liao X, Zhou Q, Kalabic J, Feagan B, Panaccione R. Maintenance Risankizumab Sustains Induction Response in Patients with Crohn's Disease in a Randomized Phase 3 Trial. J Crohns Colitis. 2024 Mar 1;18(3):416-423. doi: 10.1093/ecco-jcc/jjad168. PMID 37797293
- [Derived] Dubinsky M, Ma C, Griffith J, Crowell M, Neimark E, Kligys K, O'Connell T. Matching-Adjusted Indirect Comparison Between Risankizumab and Ustekinumab for Induction and Maintenance Treatment of Moderately to Severely Active Crohn's Disease. Adv Ther. 2023 Sep;40(9):3896-3911. doi: 10.1007/s12325-023-02546-6. Epub 2023 Jun 27. PMID 37368103
- [Derived] Loftus EV Jr, Griffith J, Neimark E, Song A, Wallace K, Nannapaneni S, Zhou J, Byrne R, Kligys K, Pang Y, Liao X, Kalabic J, Dubinsky M. Efficacy, Safety, Patient Experience, and Tolerability of Risankizumab Administered by On-Body Injector for Moderate to Severe Crohn's Disease. Adv Ther. 2023 May;40(5):2311-2325. doi: 10.1007/s12325-023-02477-2. Epub 2023 Mar 14. PMID 36917429
- [Derived] Ferrante M, Panaccione R, Baert F, Bossuyt P, Colombel JF, Danese S, Dubinsky M, Feagan BG, Hisamatsu T, Lim A, Lindsay JO, Loftus EV Jr, Panes J, Peyrin-Biroulet L, Ran Z, Rubin DT, Sandborn WJ, Schreiber S, Neimark E, Song A, Kligys K, Pang Y, Pivorunas V, Berg S, Duan WR, Huang B, Kalabic J, Liao X, Robinson A, Wallace K, D'Haens G. Risankizumab as maintenance therapy for moderately to severely active Crohn's disease: results from the multicentre, randomised, double-blind, placebo-controlled, withdrawal phase 3 FORTIFY maintenance trial. Lancet. 2022 May 28;399(10340):2031-2046. doi: 10.1016/S0140-6736(22)00466-4. PMID 35644155
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com